CLINICAL TRIAL: NCT06549439
Title: A Phase I Clinical Study on Feasibility and Toxicity of LINAC-based Flash Radiotherapy for Palliative Treatment of Skin Lesions of Malignant Melanomas
Brief Title: eFLASH for Skin Lesions of Malignant Melanomas
Acronym: Flash-Skin I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zurich Flash-Skin I
Record Dates: First submitted 2024-03-15; First posted 2024-08-12 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Melanoma
Keywords: FLASH; Radiotherapy; Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): A nominal electron energy of 9 MeV will be used for both Flash-RT and Conv-RT, which guarantees ≥ 90% dose coverage up to a depth of 2.8 cm. Shallower lesions will be treated with the same electron energy and with a bolus. In order to treat these patients, field sizes between 2x2cm2 and 10x10cm2 will be used, which can be delivered with sufficient flatness (<5%) and symmetry (<2%) by the FlashTrueBeam v2.7.5.
  Interventions: Radiation: Electron FLASH radiotherapy

INTERVENTIONS:
Radiation: Electron FLASH radiotherapy — A nominal electron energy of 9 MeV will be used for both Flash-RT and Conv-RT, which guarantees ≥ 90% dose coverage up to a depth of 2.8 cm. Shallower lesions will be treated with the same electron energy and with a bolus. In order to treat these patients, field sizes between 2x2cm2 and 10x10cm2 will be used, which can be delivered with sufficient flatness (<5%) and symmetry (<2%) by the FlashTrueBeam v2.7.5.

SUMMARY:
This prospective single center phase I trials aims to assess feasibility and safety of electron FLASH RT for treatment of melanoma skin metastases. Feasibility will be defined as FLASH delivery with an accuracy of +/-10% for each fraction, safety will be confirmed if a maximum of 2 out of 6 patients develop dose limited toxicity.

DETAILED DESCRIPTION:
Trial aim:

This prospective single center phase I trial aims to assess feasibility and safety of electron Flash RT for treatment of melanoma skin metastases. Feasibility will be defined as Flash delivery with an accuracy of ±10% for at least 10 out of 12 Flash-RT fractions and the accuracy of the total reference dose delivered (3x 9 Gy) is ±5%, safety will be confirmed if a maximum of 2 out of 6 patients develop dose-limiting toxicity.

Intervention Flash:

A nominal electron energy of 9 MeV will be used for both Flash-RT and Conv-RT, which guarantees ≥ 90% dose coverage up to a depth of 2.8 cm. Shallower lesions will be treated with the same electron energy and with a bolus. In order to treat these patients, field sizes between 2x2cm2 and 10x10cm2 will be used, which can be delivered with sufficient flatness (<5%) and symmetry (<2%) by the FlashTrueBeam v2.7.5.

Trial outline:

In the primary cohort, six patients with ≥ 1 melanoma skin lesion(s) (possible other lesions do not have to be treated) will be treated with a radiotherapy schedule of 3x 9 Gy (2x fractions/ week; α/β(3): EQD2: 64.8 Gy; α/β(10): EQD2: 42.75 Gy). A minimum of one lesion will be treated with Flash-RT (2x 9 Gy) and Conv-RT (1x 9 Gy) as experimental treatment and an optional minimum of one lesion will be treated with Conv-RT (3x 9 Gy) as "internal" control. As a consequence, also patients with a single lesion can be included into the trial. For the experimental treatment, the first two fractions will be applied with Flash-RT. Following dosimetry of these two fractions, the third fraction will be applied by Conv-RT and will be adjusted to compensate for possible lower or higher doses applied with Flash-RT before. This approach ensures that every lesion is treated with precisely a total reference dose of 27 Gy (± 5%), ultimately.

In an optional expansion cohort, up to 4 additional patients (total of n=10) will be recruited. The expansion cohort serves to further validate the primary results. The initiation of the expansion cohort requires to following three factors: 1. A maximum of 2 out of 6 patients develop DLT an no unexpected high-grade toxicity appear in the primary cohort; 2. Feasibility in the first six patients was shown (defined as Flash delivery with an accuracy of ±10% for at least 10 out of 12 Flash-RT fractions and the accuracy of the total reference dose delivered (3x 9 Gy) of ±5%); 3. No excessive duration in the recruitment of the primary cohort. Patients will be included and treated into the expansion cohort as in the primary cohort.

ELIGIBILITY:
Inclusion criteria

1. Signed study Informed Consent Form.
2. Males and females, age ≥ 18 years, no upper age limit.
3. Patients with metastatic melanoma and ≥ 1 skin/subcutaneous metastases (clearly definable in clinical examination: largest dimension of ≥ 5mm and ≤ 55 mm; ≤ 2.8 cm thickness (caliper-based measurement); volume ≤ 100ccm) with an indication for palliative radiotherapy of ≥ 1 skin/subcutaneous metastases according to the multidisciplinary tumorboard.
4. The treated lesions must be at least 5 cm apart from each other, if applicable.
5. Lesions located on the scalp can be treated.
6. ECOG 0-2. Note: Patients may receive concurrent standard of care systemic treatment.

Exclusion criteria:

1. Previous radiotherapy of the target lesions.
2. Ulcerated lesions may not be treated within the study. Patients may have ulcerated tumor lesions besides those selected for treatment within the trial.
3. Lesions, for which a homogeneous dose distribution inside the tumor D95%> 95% - D2% <107% for the PTV (acceptable deviation D90%> 80% - D2% <115%) in the treatment planning system cannot be achieved.
4. Lesions should not be located on the face. Lesions on the forehead located cranially from a line situated 1 cm above the eyebrows can be treated (=cranial of sinus frontalis).
5. Lesions should not be located directly on genitals.
6. Lesions with close proximity to air-filled cavities or air-filled, luminal organs (e.g. bowel). Close proximity is defined by intersection of the respective part of the organ at risk with the 80% isodose line of the lesion planned for radiotherapy.
7. Women who are pregnant or breast feeding.
8. Lack of safe contraception during the study, defined as: Female participants of childbearing potential and male participants with partner of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
9. Known or suspected non-compliance, drug or alcohol abuse, inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant, previous enrollment into the current study.
10. Enrollment of the investigator, his/her family members, employees and other dependent persons.
11. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Not adequately controlled HIV disease (HIV-viral load detectable).
12. Other severe comorbidities or psychiatric disorders (e.g. myocardial infraction within 6 months prior to registration, permanent cardiac arrhythmia, COPD Gold IV, schizophrenia, ongoing alcohol abuse) that would, according to the evaluation of the investigator, limit compliance with study requirement, substantially increase the risk of incurring adverse events or compromise the ability of the patient to give written informed consent.
13. History of sun hypersensitivity or photosensitive dermatoses including porphyria, systemic lupus erythematosus, Sjögren's syndrome, xeroderma pigmentosum, polymorphous light eruptions.
14. Concomitant auto-immune disease with skin lesions.
15. Concomitant use of radio-sensitizer drug.
16. Current, recent (within 10 days prior to start of study treatment), or planned participation in an experimental drug study (before end of treatment (EOT) visit).
17. Concomitant use of systemic oncological treatment for another cancer than the metastatic melanoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (Safety) | 9 months
  H0: More than of 2 out of 6 patients in the primary study cohort (n=6) develop DLT in FLASH-irradiated lesions.
  H1: A maximum of 2 out of 6 patients in the primary study cohort (n=6) develop DLT in FLASH-irradiated lesions.
Dose Accuracy (Feasibility) | 9 months
  H0: More than of 2 out of 12 Flash-RT fractions in the primary study cohort (n=6) have a dose deviation larger than ±10%.
  H1: A maximum of 2 out of 12 Flash-RT fractions in the primary study cohort (n=6) have a dose deviation larger than ±10%.

SECONDARY OUTCOMES:
Relief of Pain | 21 months
  Pain will be assessed using an analogic visual pain scale (scale 0-10; 0=no pain, 10=worst pain)
Relief of Hemorrhage | 21 months
  Hemorrhage will be visually assessed by the investigator
Local response assessment | 9 months
  Local response and control of irradiated metastases will be measured as recording of clinical response assessment including photo documentation
Late side effects | 21 months
  Late side effects "in radiation field" (≥ 3 months an within 12 months post-treatment) will be measured as recording of late adverse events (CTCAE v5.0); and comparison of Flash- and Conv-irradiated lesions

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No